CLINICAL TRIAL: NCT00639119
Title: Effect of Ropinirole Hydrochloride in Progressive Myoclonic Epilepsy of Unverricht-Lundborg Type
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: University of Turku (Other)
Responsible Party: Matti Karvonen, MD, PhD, Department of Neurology, Turku University Hospital
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: ERPME01
Record Dates: First submitted 2008-02-28; First posted 2008-03-19 (Estimated); Last update posted 2008-03-19 (Estimated); Status verified 2008-02

CONDITIONS: Unverricht-Lundborg Syndrome
MeSH Terms: conditions — Unverricht-Lundborg Syndrome | interventions — ropinirole

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Ropinirole — 8 + 8 weeks cross-over placebo controlled

SUMMARY:
The progressive myoclonus epilepsy of the Unverricht-Lundborg disease (ULD) type is an autosomal recessive disease characterized by progressive stimulus-sensitive and action-related myoclonic jerks.

The mainstay of the current treatment in myoclonic epilepsies including ULD are valproic acid and clonazepam among several other antiepileptic drugs. Unfortunately the disease may often be resistant to antiepileptic drugs leading to major reductions in daily activities and disability to walk without assistance. Therefore new treatment modalities are needed. Experimental treatments of ULD patients with dopamine agonists have relieved myoclonic symptoms. Further, in accordance with this, a recent study indicates decreased dopaminergic neurotransmission in the basal ganglia of ULD patients, determined by PET.

The purpose of this study is to investigate the effect of dopaminergic medication (ropinirole hydrochloride, Requip ®) on relieving the symptoms of ULD patients. Patients will undergo sixteen weeks intervention period. The main efficacy determinants are changes in unified myoclonus rating scale (UMRS), nerve conduction, multi-modality evoked potentials including visual evoked potential (VEP), somatosensory evoked potential (SSEP) and brainstem auditory evoked potential (BAEP), blink reflex habituation and electroencephalography (EEG). Tolerability and the safety of the medication are determined. The study setting is placebo controlled, crossover, two-group and double blind study.

ELIGIBILITY:
Inclusion Criteria:

* Unverricht-Lundborg Syndrome

Exclusion Criteria:

* Pregnancy
* Intolerability to ropinirole hydrochloride
* Mental illness

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2007-08; Primary Completion 2008-08 (Estimated)

PRIMARY OUTCOMES:
Unified myoclonus rating scale | 3

CONTACTS AND LOCATIONS:
Locations (1):
- Turku university central hospital, Department of neurology, Turku, Finland